CLINICAL TRIAL: NCT05189379
Title: Targeted Extinction of Drug Cues During Sleep - Olfactory Cue Reactivity Task
Acronym: TEDDS_OCRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: tedds_ocrt_1
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Heavy Drinking
Keywords: Cue Reactivity Task; Heavy Drinking; Olfactory Cue Reactivity Task
MeSH Terms: interventions — 2-methyltetrahydrofuran-3-one; Beer; Wine

STUDY DESIGN:
Intervention Model Description: A two group study is constructed with the sole intention to balance the amount of participants who would undergo the same experiment with a different order. Half of the participants will receive odour based Cue Reactivity Task first, other half will complete the image based Cue Reactivity Task first.
  Before the MRI screening participants would be asked about their preference between beer, wine and schnapps then during the odour based Cue Reactivity Task only their preferred beverage odour would be delivered.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olfaction First (Experimental): Participants assigned to this arm will undergo the experiment in the following order: Odour based Cue Reactivity Task, Monetary Incentive Delay Task, Image based Cue Reactivity Task
  Interventions: Other: Non-Alcoholic Odour; Other: Alcoholic Odour; Other: Non-Alcoholic Images; Other: Alcoholic Images
- Image First (Experimental): Participants assigned to this arm will undergo the experiment in the following order: Image based Cue Reactivity Task, Monetary Incentive Delay Task, Odour based Cue Reactivity Task
  Interventions: Other: Non-Alcoholic Odour; Other: Alcoholic Odour; Other: Non-Alcoholic Images; Other: Alcoholic Images

INTERVENTIONS:
Other: Non-Alcoholic Odour — A chemical used in fragrances and flavouring with a smell close to a nutty, buttery structure. Used as a 1:100 deionised water dilution.
  Other Names: Coffee furanone; 2-Methyltetrahydrofuran-3-one
Other: Alcoholic Odour — Alcoholic beverage beer / Alcoholic beverage red wine / Alcoholic beverage brandy / The type of the Alcoholic Odour intervention will be presented in a participant-preference basis.
  Other Names: Beer; Wine; Schnapps
Other: Non-Alcoholic Images — Images of non-alcoholic items, namely; broom, duster, clothing iron, lightbulb, mat, mulch, penlight, rack, rock, kitchen scissors, trough, vent are presented in parallel with the non-alcoholic odour
Other: Alcoholic Images — Images of alcoholic items, namely, beer, wine, schnapps are presented in parallel with the alcoholic odour

SUMMARY:
The study aims to utilise olfactory stimulation in addition to the visual stimulation in cue reactivity tasks to enhance precision in measuring alcohol based cues in individuals diagnosed with heavy drinking. The study consists of one cue reactivity task with visual stimuli, another cue reactivity task with matching odour/visual stimuli and lastly a monetary incentive delay task.

DETAILED DESCRIPTION:
The intention of the study is to enhance the measurement precision in image-based cue reactivity task by introducing a new level of stimuli in the form of odours. During the course of the functional Magnetic Resonance Imaging (fMRI) screening, participants are required to finish three tasks, namely; odour-based cue reactivity task (OCRT), image-based cue reactivity task(ICRT) and monetary incentive delay task (MID).

Participants will be randomly divided into two groups, one group will receive tasks in the following order: OCRT-MID-ICRT and the other group will receive them in the following order: ICRT-MID-OCRT. With this, the habituation effect from receiving odours during OCRT is expected to be balanced.

ELIGIBILITY:
Inclusion Criteria:

* An Heavy Drinking diagnosis, confirmed by Alcohol Use Disorders Identification Test
* Ability to provide fully informed consent and to use self-rating scales in fMRI
* Understanding of the German language

Exclusion Criteria:

* Severe mental or physical illnesses
* Insomnia
* Any metal parts and pieces in the body
* Claustrophobia; fear of confined spaces

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Change in Blood Oxygen Level Dependent (BOLD) signal within selected Regions of Interest (ROI) | Once during the fMRI experiment
  Change in brain activation in the form of BOLD signals within 3 groups of ROIs:
  * Memory related ROIs: Hippocampus, Dorsolateral Prefrontal Cortex
  * Cognitive Control related ROIs: Anterior Cingulate Cortex, Ventrolateral Prefrontal Cortex
  * Reward related ROIs: Striatum (ventral and dorsal) and Insula
Odour based cue reactivity task | Once during the fMRI screening
  A cue reactivity task based on the odours and images of alcoholic and non-alcoholic items. Adapted from Vollstädt-Klein et al., 2011.
  Subjects are presented with odours and images of alcoholic (beer, wine, schnapps) and non-alcoholic (odour: 2-Methyltetrahydrofuran-3-one / images: broom, duster, clothing iron, lightbulb, mat, mulch, penlight, rack, rock, kitchen scissors, trough, vent) items during an fMRI session in blocks. For non-alcoholic items, in each block 5 images from the same stimuli group are presented with the non-alcoholic odour. For alcoholic items, in each block there are 5 images from the selected stimuli group with the congruent odour.
  After each block subjects are asked to rate their liking and wanting towards the items that have been presented to them in two 1-5 scales. Blocks are pseudorandomised to maximise balance between groups and minimise the effect of habituation.
  Minimum 1: "not at all", maximum 5: "very much".
Image based cue reactivity task | Once during the fMRI screening
  A cue reactivity task based on the images of alcoholic and non-alcoholic items. Adapted from Vollstädt-Klein et al., 2011.
  Subjects are presented with images of the alcoholic (beer, wine, schnapps) and the non-alcoholic (broom, duster, clothing iron, lightbulb, mat, mulch, penlight, rack, rock, kitchen scissors, trough, vent) items during an fMRI session in blocks. In each block there are 5 images from the same stimuli group. After each block subjects are asked to rate their liking and wanting towards the items that have been presented to them in two 1-5 scales. Blocks are pseudorandomised to maximise balance between groups and minimise the effect of habituation.
  Minimum 1: "not at all", maximum 5: "very much".
Monetary incentive delay task | Once during the fMRI screening
  A task to invoke reward based activations in the subjects. Adapted from Kirsch et al., 2003.
  Subjects are presented 3 different stimulus conditions, each linked either to a positive monetary reward (a vertically oriented arrow pointing upward), a positive verbal feedback (a vertically oriented double-sided arrow) or a neutral no reward or feedback (a horizontally oriented double-sided arrow). After presentation of the two positive stimuli types, a flashing screen is presented and during the flashing screen if the subjects can press the button fast enough they will either win 1€ or they will be shown a positive verbal feedback depending on the positive stimuli type. The negative stimuli is followed by a 3 second black screen to include a control condition. Each stimulus condition is presented 10 times in a pseudorandom schedule with no more than two equal conditions in succession. The inter-trial interval randomly varies between 6-9 seconds.

SECONDARY OUTCOMES:
Psychomotor Vigilance Test (Roach et al. 2006) | Once before the fMRI screening
  Task measuring the objective vigilance of subjects. To distinguish vigilance between the wake and the sleep conditions, following measures will be compared: Median reaction speed (1/reaction time) and percentage of lapses (number of lapses divided by the number of all valid stimuli, excluding false starts. Lapse >= 500 ms, false start < 100ms). The task is prepared in JsPsych, and administered with using a tablet connected to internet. Participant data is securely stored in an encrypted server.
Stanford Sleepiness Scale (Hoddes et al. 1973) | Once before the fMRI screening
  Test measuring current level of alertness of subjects on a seven point scale. A high test score indicates a high level of sleepiness and conversely a low test score yields a low level of sleepiness. Test scores will be utilized as a pre-measurement alertness indicator for participants. The task is prepared in JsPsych, and administered with using a tablet connected to internet. Participant data is securely stored in an encrypted server.
Alcohol Urge Questionnaire (Bohn et al. 1995) | Once before the fMRI screening
  Questionnaire on self-assessment of current craving of subjects. Consists of 8 items on a Likert-type scale from 1-7 where higher scores represent stronger alcohol urges. The task is prepared in JsPsych, and administered with using a tablet connected to internet. Participant data is securely stored in an encrypted server.
Sniffin' Sticks Test (Burghardt®, Wedel, Germany)(Hummel et al., 1997) | Once before the fMRI screening
  A psychophysical test that is developed for assessing individuals reactions to the olfactory stimuli (Hummel et al., 1997). The 12-stick test from Burghardt is chosen for the study and it consists of identifying one of the four items that are presented with each of the twelve odourant sticks. At the end, with the aid of the identification score, the participant's olfaction capability is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon B Feld, Dr, Principal Investigator — ZI Mannheim, Department of Clinical Psychology, RG Psychology and Neurobiology of Sleep and Memory
Locations (1):
- Zentralinstitut für Seelische Gesundheit Mannheim, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No
Due to data protection rules, individual data cannot be shared. Cumulated data on the group level can be made available for meta-analyses on request.

REFERENCES:
- [Background] Vollstadt-Klein S, Loeber S, Kirsch M, Bach P, Richter A, Buhler M, von der Goltz C, Hermann D, Mann K, Kiefer F. Effects of cue-exposure treatment on neural cue reactivity in alcohol dependence: a randomized trial. Biol Psychiatry. 2011 Jun 1;69(11):1060-6. doi: 10.1016/j.biopsych.2010.12.016. Epub 2011 Feb 3. PMID 21292243
- [Background] Roach GD, Dawson D, Lamond N. Can a shorter psychomotor vigilance task be used as a reasonable substitute for the ten-minute psychomotor vigilance task? Chronobiol Int. 2006;23(6):1379-87. doi: 10.1080/07420520601067931. PMID 17190720
- [Background] Hoddes E, Zarcone V, Smythe H, Phillips R, Dement WC. Quantification of sleepiness: a new approach. Psychophysiology. 1973 Jul;10(4):431-6. doi: 10.1111/j.1469-8986.1973.tb00801.x. No abstract available. PMID 4719486
- [Background] Bohn MJ, Krahn DD, Staehler BA. Development and initial validation of a measure of drinking urges in abstinent alcoholics. Alcohol Clin Exp Res. 1995 Jun;19(3):600-6. doi: 10.1111/j.1530-0277.1995.tb01554.x. PMID 7573780
- [Background] Hummel T, Sekinger B, Wolf SR, Pauli E, Kobal G. 'Sniffin' sticks': olfactory performance assessed by the combined testing of odor identification, odor discrimination and olfactory threshold. Chem Senses. 1997 Feb;22(1):39-52. doi: 10.1093/chemse/22.1.39. PMID 9056084
- [Background] Kirsch P, Schienle A, Stark R, Sammer G, Blecker C, Walter B, Ott U, Burkart J, Vaitl D. Anticipation of reward in a nonaversive differential conditioning paradigm and the brain reward system: an event-related fMRI study. Neuroimage. 2003 Oct;20(2):1086-95. doi: 10.1016/S1053-8119(03)00381-1. PMID 14568478